CLINICAL TRIAL: NCT04653220
Title: Metabolic Response Evaluation of Low-sugar Snack Bars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2019/00861
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Pre Diabetes; Diabetes; Obesity
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized crossover study
Who Masked: Participant
Masking Description: Participant is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control 1 (Other): Glucose 25g
  Interventions: Other: Control 1
- Control 2 (Other): Glucose 25g
  Interventions: Other: Control 2
- Standard Crokao (Experimental): Commercially available snack bar
  Interventions: Other: Standard Crokao
- Low sugar variant 1 (Experimental): Low sugar snack bar with sticky rice
  Interventions: Other: Low sugar variant 1
- Low sugar variant 2 (Experimental): Low sugar snack bar with promitor
  Interventions: Other: Low sugar variant 2
- Low sugar variant 3 (Experimental): Low sugar snack bar with inulin
  Interventions: Other: Low sugar variant 3
- Low sugar variant 4 (Experimental): Low sugar snack bar with yellow soy
  Interventions: Other: Low sugar variant 4
- Low sugar variant 5 (Experimental): Low sugar snack bar with rice syrup
  Interventions: Other: Low sugar variant 5

INTERVENTIONS:
Other: Control 1 — 25g glucose dissolve in 250ml of water
  Arms: Control 1
Other: Control 2 — 25g glucose dissolve in 250ml of water
  Arms: Control 2
Other: Standard Crokao — Standard Crokao containing 25g of available carbohydrate
  Arms: Standard Crokao
Other: Low sugar variant 1 — Low sugar variant 1 containing 25g of available carbohydrate
  Arms: Low sugar variant 1
Other: Low sugar variant 2 — Low sugar variant 2 containing 25g of available carbohydrate
  Arms: Low sugar variant 2
Other: Low sugar variant 3 — Low sugar variant 3 containing 25g of available carbohydrate
  Arms: Low sugar variant 3
Other: Low sugar variant 4 — Low sugar variant 4 containing 25g of available carbohydrate
  Arms: Low sugar variant 4
Other: Low sugar variant 5 — Low sugar variant 5 containing 25g of available carbohydrate
  Arms: Low sugar variant 5

SUMMARY:
To determine the post-prandial metabolic response and biomarker response, following the consumption of newly developed low glycaemic index (GI) snack bars. The snack bars are formulated with different combinations and ratios of ingredients and food structures. The low sugar products maintaining glucose homeostasis and preventing metabolic problems may have commercial potential as a novel functional ingredient in a variety of fields, including nutrition, medicine, and agriculture.

DETAILED DESCRIPTION:
In this study we will study and compare the postprandial metabolic response of 5 snack bar variants, 1 control product and 2 glucose (25g) reference drinks. The study will have a total of 8 test sessions in a non-blinded, crossover design. Online computer software will be used for simple randomization of the sequence of the 8 treatments (http://www.randomizer.org/).The 5 snack bars variants will be similar in macronutrient composition but will differ in the source of carbohydrate, fibre and protein (rice, bamboo, inulin, soy, promitor). They will be compared to a visually similar control product (crokao) that is higher in sugar. The reference drink will be anhydrous glucose (25g) dissolved in 250 ml of water.Study population: 15-20 participants will be recruited from each of the following ethnicities: Chinese, Indian and Caucasian. During the screening session, participants will receive an informed consent form and given ample time to go through it and rectify any queries they have with the researcher. The number of test sessions will be discussed between the researcher and the participants, depending on the volunteer's schedule. If they decide to take part in the study, they will be asked to sign the informed consent form. They will then be asked to complete a screening questionnaire and subsequently baseline measurements including anthropometric measurements, blood pressure, and fasting blood glucose will be collected from each participant in order to determine their eligibility. The screening questionnaire will include demographic, general health details, and physical activity level. This information will be used to determine whether the participant is eligible for the study, as well as to check for any possible confounders that may influence the study outcomes. Anthropometric measurements: Body weight and body composition will be measured using bioelectrical impedance analysis (Tanita scale). Height will be measured using a stadiometer in order to calculate participants' BMI. Waist circumference will be measured at the minimum circumference between the iliac crest and the rib cage and hip circumference will be measured at the maximum protuberance of the buttocks. Blood pressure will be measured using an Omron blood pressure monitor (Model HEM-907) at baseline. Participants will be seated for five minutes before blood pressure is measured. Measurements will be taken in duplicate and the averaged results will be recorded.

Study protocol: The day before a test day, participants will be encouraged to consume their usual diet and avoid alcohol consumption and participating in vigorous exercise. On test days, participants will arrive at the laboratory after an overnight fast of 10 h. Upon arrival, participants will be asked to void, and have their weight and body fat assessed with a Tanita scale. After that, participants will enter the clinical suit and rest for 15 min before a blood catheter is inserted in the antecubital vein of the arm. After the blood catheter is inserted, participants will rest for 15 min, before two baseline blood sample (6 mL) are taken 10 minutes apart (-10 min and 0 min). Immediately after the second sample, participants will be served a test food that has to be consumed within 15 min. Subsequently blood samples (6mL) are obtained at 15, 30, 45, 60, 90,120, 180 and 240min. Appetite sensations (e.g. hunger, fullness, desire-to-eat etc.) will also be measured using questionnaires at similar time points when blood samples are taken. Subjects will be asked to rate their appetite sensations on a 100 mm visual analogue scale (VAS). After each session, the blood catheter will be removed. The participants will leave the laboratory and they will be asked to keep a food diary of what they eat for the remaining day. Participants will return until all test foods are consumed. During the entire test session, the subject will have to stay rested and in the laboratory. Television and a workspace will be provided to the subject.Blood samples will be will analysed for METABOLIC RESPONSE (glucose, insulin, Triglycerides, NEFA, GLP-1 and ghrelin). A 100 uL aliquot of blood during the first blood sample collection (T = -10min) will be obtained from each participant on the first day of treatment (thus only once) for baseline metabolomics profiling.A stool sample from each participant will be obtained to perform the following on the microbiome: DNA extraction, library prep, 16S and shotgun (whole genome) sequencing, and demultiplexing of genomic data. The stool sample will be collected between the screening session and the last test session (time of collection will not influence the sample analysis). The participant will be encouraged to collect the stool sample during one of the sessions at the research centre to eliminate transport of the sample.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 21-65 years
* Chinese, Indian and Caucasian Ethnicity
* Body mass index between 18.5 - 25.5 kg/m2
* Fasting blood glucose <7.0 mmol/L
* Normal blood pressure (<140/90 mmHg)
* In general good health

Exclusion Criteria:

* Smoking
* Partake in sports at a high competitive and/or endurance levels
* Intentionally restrict food intakeHave known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Have poor veins impeding venous access and have any history of severe vasovagal syncope (blackouts or near faints) following blood draws
* Have metabolic diseases (such as diabetes, hypertension, etc.)
* have medical conditions and/or taking medications known to affect glycemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* Have any major organ dysfunction (e.g. cardiovascular, respiratory, hepatic, renal, gastrointestinal) that may influence taste, olfaction, appetite, digestion, metabolism, absorption or elimination of test foods, nutraceutical or drug,
* Have any severe food allergy or food intolerance
* Having active Tuberculosis (TB) or currently receiving treatment for TB
* Have any known Chronic Infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Are a member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Concurrent participation in a study that might affect the outcomes of the current study

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All healthy male subjects
Enrollment: 48 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Change in postprandial blood glucose over 240 minutes period | 240 minutes
  Venous Blood obtained through canula, analysed using Beckman Coulter analyser.

SECONDARY OUTCOMES:
Change in postprandial plasma insulin over 240 minutes period | 240 minutes
  Venous blood obtain through cannula, analysed using Beckman Coulter analyser.
Change in postprandial plasma triglycerides over 240 minutes period | 240 minutes
  Venous blood obtain through cannula, analysed using Beckman Coulter analyser.
Change in postprandial plasma non esterified fatty acids over 240 minutes period | 240 minutes
  Venous blood obtain through cannula, analysed using chemistry analyser.
Change in postprandial plasma active ghrelin over 240 minutes period | 240 minutes
  Venous blood obtain through cannula, analysed using ELISA analyser.
Change in postprandial plasma active GLP-1 over 240 minutes period | 240 minutes
  Venous blood obtain through cannula, analysed using ELISA analyser.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore